CLINICAL TRIAL: NCT05895175
Title: Assessing the Evolution of Maternal and Paternal-fetus Attachment in Couples Conceiving Through Egg Donation
Brief Title: Evolution of Maternal and Paternal-fetus Attachment in Egg Donation
Status: Completed | Type: Observational
Sponsor: Fundación IVI (Other)
Responsible Party: Sponsor
Other Study IDs: 2112-ROM-108-MF
Record Dates: First submitted 2023-05-11; First posted 2023-06-08 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2023-05

CONDITIONS: Perinatal Disorder
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DONATED GAMETE GROUP: couples who got pregnant through egg donation (with their own semen)
  Interventions: Other: Questionnaires
- OWN GAMETE GROUP: couples who got pregnant through standard IVF treatment, with their own gametes
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Questionnaires

SUMMARY:
Recently, many families have been formed through gamete donation, a reproductive treatment where the ensuing children do not share a genetic link with either parents. However, despite such an increase, little is known about the parent-child relationship. Indeed, only two longitudinal studies have provided scientific background about family functioning in gamete donation. These studies showed that in egg donation families, the parent-child relationship was normal for parenting, parent psychological health, and child adjustment.

A more recent study evaluated mother-infant interaction in egg donation families comparing them with those created through IVF with their own gametes. Data collected showed that in egg donation families the mother-infant relationship quality appeared to be less optimal. Mothers were less interactive and stimulating, and infants showed lower involvement and less responsiveness with respect to their mothers Overall, the evidence suggests that women conceiving through egg donation likely require a variable period of adaptation to parenting. Here, the investigators aim to evaluate this interaction at an earlier stage, that is during the gestation. The specific bond that parents develop towards the fetus during pregnancy is called "parental-fetus attachment". Previous studies showed that the quality of the parental-fetus attachment is predictive of the quality of the postnatal parent-infant relationship and the child development The purpose is to evaluate whether the lack of genetic link with their offspring could undermine the parental attachment to the fetus, comparing couples conceiving through egg donation with those who get pregnant through a standard IVF treatment with their own gametes. No studies have been performed so far on this matter.

To assess the mother-father fetus attachment, the investigators will administer standardized and validated questionnaires to couples undergoing IVF with their own gametes, or egg donation cycles. For women, the investigators will use the Maternal Antenatal Attachment Scale . For men, the investigators will use the Paternal Antenatal Attachment Scale (PAAS-IT) . Furthermore, to also assess the emotional status of both partners, the investigators will use the Matthey Generic Mood Questionnaire .

Seeing that in the general population the maternal-fetal attachment level increases once women have completed the principal prenatal genetic screenings (like NIPT, CVS or amnio) and once they start perceiving the fetal movements, the investigators will administer the same questionnaire twice: between the 19-23 weeks and between the 28-32 weeks of gestation. This approach will enable monitoring of the evolution of the maternal and paternal fetal attachment at relevant gestational time-points.

As a result of the knowledge gathered from this study, the investigators will be able to develop a specific intervention strategy to promote this fundamental process for egg donation families.

ELIGIBILITY:
DONATED GAMETE GROUP

Inclusion criteria:

* getting pregnant through an egg donation program
* Own semen
* Native language must be English or Italian

Exclusion criteria:

* Patients failing to consent to be recontacted for research purpose.
* Patients who are taking psychotropic drugs
* Patients who got pregnant through sperm or embryo donation

OWN GAMETE GROUP

Inclusion criteria:

* getting pregnant through a standard IVF treatment with own gametes
* Native language must be English or Italian

Exclusion criteria:

* Patients failing to consent to be recontacted for research purpose.
* Patients who are taking psychotropic drugs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The reference population includes all couples who have become pregnant in the selected IVI RMA clinics , through egg donation or standard IVF treatment, being the woman 40 years old or above, with no other specific indications (except individuals taking psychotropic drugs). Their native language must be English or Italian.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
validated questionnaire to assess the change of maternal fetus attachment (MAAS) | between 19-23 gestational weeks and follow up between 28-32 weeks of gestation
  The MAAS total score is calculated by the sum of all item of the questionnaire, and the subscales score (quality and intensity of the attachment) are calculated through the sum of the rate of each item that is included in that scale. Scoring is 1-5, with 5 high attachment
validated questionnaire to assess the change of Paternal fetus attachment (PAAS) | between 19-23 gestational weeks and follow up between 28-32 weeks of gestation
  The PAAS total score is calculated by the sum of all item of the questionnaire, and the subscales score (quality and intensity of the attachment) are calculated through the sum of the rate of each item that is included in that scale. Scoring is 1-5, with 5 high attachment
questionnaire to explore the change of the Emotional status (Anxiety or depression feelings) during pregnancy (MGMQ) | between 19-23 gestational weeks and follow up between 28-32 weeks of gestation
  The MGMQ provideds a screen positive / negative classification of emotional distress

CONTACTS AND LOCATIONS:
Locations (3):
- IVI Roma, Roma, Italy
- IVI Foundation, Valencia, Spain
- IVI London, London, United Kingdom